CLINICAL TRIAL: NCT06881407
Title: Effect of a Humanoid Robot With Virtual Reality Games to Train Arm Function in Children With Cerebral Palsy - THRIVE Trial
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Yuping Chen, Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H23116; 90IFST0009 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2025-02-27; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Virtual Reality; Humanoid Robot; Home-based Intervention; Arm Function
MeSH Terms: conditions — Cerebral Palsy | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE (Combination of Virtual Reality and Humanoid Robot) (Experimental): Participants will receive the home-based intervention using the combination of virtual reality and a humanoid robot, "who" serves as a cheerleader and coach, for 8 weeks. During each week, participants will need to exercise 3 sessions per week, for around 60 minutes per session.
  Interventions: Device: Robot; Device: Virtual Reality
- Virtual Reality Alone (Active Comparator): Participants will receive the home-based virtual reality intervention for 8 weeks. During each week, participants will need to exercise 3 sessions per week, for around 60 minutes per session.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Robot — This robot will serve as a cheerleader and coach to provide encouragement and feedback.
  Other Names: Humanoid Robot
  Arms: THRIVE (Combination of Virtual Reality and Humanoid Robot)
Device: Virtual Reality — Our developed Super Pop VR system will be used to provide virtual reality intervention.
  Other Names: VR

SUMMARY:
About 60% of children with cerebral palsy (CP) have impaired arm function. Improving arm function requires hundreds of repetitions per day, which is impossible in a single clinical visit. Thus, therapeutic exercises should be sustained in the home environment; however, the compliance in performing home exercise is low due to poor motivation, boredom, and forgetfulness. A better home program is needed. The objective of this project is to examine the effect of our developed "THRIVE" system (Therapeutic Humanoid Robot In Virtual Environment: the combination of robot with virtual reality games), which can provide a motivating and tailored upper-extremity intervention program with instant feedback, to improve arm function in children with CP at their home. The investigators believe the newly developed "THRIVE" system can increase children's engagement and motivation in home exercises as the robot is their playmate to demonstrate and correct their movements. The investigators will also interview parents and children with CP to understand their impression of using technology at home to shape the intervention. The expected outcome is that children with CP receiving "THRIVE" will improve their arm function more and have better engagement than those who receive VR alone immediately after intervention and at follow-up. The long-term goal is to have the "THRIVE" system be the optimal home exercise platform as it can provide challenging but motivating exercises to improve children's arm function while assisting parents in supervising their children with CP to complete home exercises.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are between the ages of 5 and 21 years;
2. diagnosed with spastic CP;
3. have a manual ability classification system (MACs) level I-III;
4. able to sit with trunk supported;
5. are able to reach forward for more than half of their arm length;
6. are able to comprehend and complete a three-steps commands;
7. are able to see a TV screen (with or without corrected vision); and
8. their primary caregiver is willing to follow the desired intervention dosing and all evaluation measurements.

Exclusion Criteria:

1. they have received surgery or botulinum toxin type A injection in the training arm within the preceding 4 months or are scheduled to receive it during the planned intervention period, or
2. if they have a severe attention deficit or uncontrolled epilepsy, which may possibly be triggered by the light or sound of the video games.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Reaching kinematics | Baseline, at 9th week, and at 13th week.
  Reaching kinematics will be assessed while the child is interacting with Super Pop VR, wherein virtual bubbles are projected onto the standard projecting screen in randomly dispersed locations using the Kinect system. Three testing bubbles will be situated in the location where children need to reach about arm length overhead at 180°, 135°, and 90° of shoulder abduction, with instructions for children to reach in two conditions: (1) as fast as possible and (2) as accurate as possible. Children's reaching kinematics will also be assessed while playing the real-life functional activity using the Kinect camera. All children will be seated in an adjustable chair with a testing table in front of them at waist height with trunk support. Data will be collected for a minimum of six reaches for each direction of virtual and real-life tasks.
Standardized fine motor assessment score | Baseline, at 9th week, and at 13th week.
  The fine motor domain of the Peabody Developmental Motor Scales, 2nd edition (PDMS-2), including grasping and visual-motor integration will be used.
Daily use of affected hand | Baseline, at 9th week, and at 13th week.
  Daily use of affected hand will be evaluated using the Revised Pediatric Motor Activity Log (R-PMAL), which is filled out by primary caregivers about how often and how well their child uses the affected arm in daily activities.

SECONDARY OUTCOMES:
Muscle strength | Baseline, at 9th week, and at 13th week.
  Muscle strength of shoulder flexion, extension, abductor, adduction, external rotation, internal rotation, elbow flexion and extension, and wrist flexion and extension will be measured using a hand-held dynamometer prior to and after intervention as well as at follow-up.
Range of Motion (ROM) | Baseline, at 9th week, and at 13th week.
  ROM of shoulder flexion, extension, abduction, adduction, external rotation, internal rotation, elbow flexion and extension, and wrist flexion and extension will be measured using a standardized goniometer.
Spasticity | Baseline, at 9th week, and at 13th week.
  Spasticity of shoulder flexion, extension, abduction, adduction, external rotation, internal rotation, elbow flexion and extension, and wrist flexion and extension will also be measured using the Modified Ashworth Scale. It contains a scale of 0 to 4 with 0 as no spasticity to 4 as rigid in flexion or extension.

OTHER OUTCOMES:
Qualitative outcome | Baseline, at 9th week, and at 13th week.
  Researcher will conduct semi-structured interview to explore the parents' and children's expectations (pre-intervention) and perceptions (post-intervention and follow-up) as well as knowledge (all 3 timepoints) about the technology we used to conduct the intervention and about the barriers and facilitators to have parents implement the technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Real user therapy assessment and outcome data and intervention log will be possibility shared to a NIH-funded open video-based data-sharing system for developmental science (i.e., Databrary). Databrary is one of the first large-scale repository for sharing video data and related information so the researchers can share and view on another's databases to promote greater transparency and peer oversight into data collection methods and measurement. All the videos collected through Kinect camera during interventions and evaluations will be de-identified first before sharing to Databrary. A new written permission will be obtained from the parents of children with CP before initiating the data sharing process. PI, Co-PI, and research team members will contact the parents to explain the purpose of data sharing. If parents show their initial agreement, a de-identified video will send it to the parents for review before uploading and sharing to Databrary.
Supporting Information: CSR
Time Frame: 9/1/2027 - after the data collection is completed and data have been analyzed and disseminated. Data will be available until 12/31/2035.
Access Criteria: Reserachers who also sign up to participate in datasharing in Databrary.

REFERENCES:
- [Background] Chen Y, Garcia-Vergara S, Howard AM. Effect of feedback from a socially interactive humanoid robot on reaching kinematics in children with and without cerebral palsy: A pilot study. Dev Neurorehabil. 2018 Nov;21(8):490-496. doi: 10.1080/17518423.2017.1360962. Epub 2017 Aug 17. PMID 28816558
- [Background] Howard A, Chen Y, Park CH. From Autism Spectrum Disorder to Cerebral Palsy: State-of-the-Art in Pediatric Therapy Robots. In Encyclopedia of Medical Robotics, J. P. Desai (Ed.), World Scientific Publishing Company, 2018, pp241-261
- [Background] Chen YP, Howard AM. Effects of robotic therapy on upper-extremity function in children with cerebral palsy: A systematic review. Dev Neurorehabil. 2016;19(1):64-71. doi: 10.3109/17518423.2014.899648. Epub 2014 Apr 11. PMID 24724587
- [Background] Chen Y, Fanchiang HD, Howard A. Effectiveness of Virtual Reality in Children With Cerebral Palsy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2018 Jan 1;98(1):63-77. doi: 10.1093/ptj/pzx107. PMID 29088476